CLINICAL TRIAL: NCT06985680
Title: Exploring the Impact of Artificial Intelligence-Based Health Education on Self-Efficacy, Self-Care Behaviors, and Glycemic Control in Diabetic Patients
Brief Title: Diabetic Patients,Self-Efficacy,Self-Care Behaviors,Artificial Intelligence-Based
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chia-Tzu Line (Other)
Responsible Party: Sponsor-Investigator, Chia-Tzu Line, head nurse, WeiGong Memorial Hospital
Organization: WeiGong Memorial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WeiGongMemorial
Record Dates: First submitted 2024-03-10; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Patients,Self-Care,Artificial Intelligence-Based,Self-Efficacy; Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LINE@ Diabetes Health Education Chatbot (Other): The research involves the application of the "Diabetes Smart Helper" LINE@ Diabetes Health Education Chatbot for intervention measures. This application includes AI automatic message responses and provides push notifications of diabetes-related medical and healthcare knowledge to ensure that the public receives accurate medical information (Chinese Diabetes Health Education Association, 2021).
  Interventions: Behavioral: LINE@ Diabetes Health Education Chatbot

INTERVENTIONS:
Behavioral: LINE@ Diabetes Health Education Chatbot — Upon opening the LINE application, the research subjects need to enter "Diabetes Smart Helper" in the LINE@ Diabetes Health Education Chatbot. Once added to the program, the LINE interface will directly display six small windows for diabetes symptoms/complications, diet, medication, exercise, mental health, and others, facilitating self-selection by users.

SUMMARY:
This study employed an experimental research design using a randomized controlled trial methodology. Group allocation was performed randomly by generating serial numbers through a computer. Participants were then randomly assigned to either the experimental or control group by placing the serial numbers into opaque envelopes and selecting envelopes in random order as patients arrived for appointments.

The experimental group received conventional face-to-face education in addition to participating in the "Diabetes Smart Assistant" Line@ diabetes education robot program. Education was delivered individually in a one-on-one manner. Researchers spent 15 minutes instructing participants on the operation and usage of the Line@ diabetes education robot program, followed by educational content delivery. Educational sessions lasted for 30 minutes on the day of enrollment, and 15 minutes each at the 3rd and 6th months of enrollment, totaling three one-on-one educational sessions. Additionally, participants received telephone consultations for follow-up during the enrollment period. Telephone education sessions were conducted in the first week of enrollment, the second month, and the fourth month, each lasting 10 minutes, totaling three sessions.

The control group received routine education and had follow-up visits every three months for one-on-one education. Data collection for both groups occurred at the time of enrollment, and at the 3rd and 6th months of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes by a physician and enrolled as a patient in the Diabetes Collaborative Care Network.
2. Aged 18 years or older.
3. Owns a smartphone and agrees to join the "Diabetes Smart Helper" LINE@ Diabetes Health Education Chatbot application.
4. HbA1c level greater than 7.0% (as referenced in Changsieng et al., 2023; Selçuk-Tosun & Zincir, 2019).

Exclusion Criteria:

1. Patients undergoing hemodialysis or peritoneal dialysis.
2. Patients diagnosed with mental illness.
3. Illiterate patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
The Chinese Version Diabetes Management Self-Efficacy Scale | 6 months.
  This study employs the Chinese Version Diabetes Management Self-Efficacy Scale (C-DMSES) developed by S. F. Wu et al. (2008) for assessment. The scale covers nutrition (9 items), exercise and weight control (4 items), medication management (3 items), and blood glucose and foot care (4 items). Scoring is based on an 11-point Likert scale, where 10 points indicate "very confident" and 0 points indicate "not confident at all." The total score ranges from 0 to 200, with higher scores indicating stronger self-efficacy, meaning that patients have greater confidence in performing diabetes self-care behaviors such as blood glucose monitoring, dietary management, control, and medication adherence. This scale is used for patients with type 2 diabetes in Taiwan, and the internal consistency reliability of the four subscales is as follows: dietary self-efficacy (α = .93), adherence to medical advice self-efficacy (α = .79), exercise and weight control self-efficacy (α = .81), and blood glucose mo
The Summary of Diabetes Self-Care Activities | 6 months.
  The Summary of Diabetes Self-Care Activities (SDSCA) published by Toobert et al. (2000) was used, which includes 25 questions covering six aspects, including diet, exercise, self-monitoring of blood glucose, smoking, self-care behavior counseling, and medication. The questionnaire was modified by Qiu (2002) to measure the self-care behavior of diabetes in Chinese. There are 10 structured questions, including foot care (3 questions), diet (2 questions), exercise (2 questions), medication (2 questions) and blood sugar monitoring (1 question). This scale monitors the daily self-care of diabetes in the past 7 days. The second question is a reverse question, and the other questions are scored in a positive way. The 7-day frequency method is used for calculation. The questionnaire scale is calculated from 0 to 7 points. Each question has a maximum score of 7 points and a minimum score of 0. For example, if the questions in the questionnaire are completed for 1 day, it represents 1 point, an
blood glucose control | 6 months.
  This study is based on the 2022 Clinical Care Guidelines for Type 2 Diabetes. Blood sugar control indicators include blood sugar level before meals, blood sugar level 2 hours after meals, and HbA1c value. It is recommended that good blood sugar control indicators for patients with type 2 diabetes are blood sugar level before meals maintained at 80-130 mg/dl, blood sugar level 2 hours after meals maintained at 80-160 mg/dl, and HbA1c value < 7.0% (Diabetes Society of the Republic of China, 2022). The above test values are from the medical records of the subjects.
  The testing equipment used by the hospital in this case has passed ISO 1589:2012, with the certification number 1575, and meets the relevant standards. According to the requirements of the National Health Insurance Diabetes Medical Benefit Improvement Program, diabetic patients must undergo a blood test every 3 months. Patients must complete the blood test 3 to 7 days before outpatient consultation. The blood draw time of th

CONTACTS AND LOCATIONS:
Overall Officials: chia-tzu lin, Principal Investigator — not related
Locations (1):
- Wei Gong Memorial Hospital, Taiwan, Toufen City, China

IPD SHARING:
Plan to Share IPD: No